CLINICAL TRIAL: NCT04099394
Title: Randomized Controlled Trial of Group-Based Exercise and Behavioral Health Skills Training for Older Adults with Painful Knee Osteoarthritis
Brief Title: Pain & Aging: Combined Interventions for Fitness in the Community Study
Acronym: PACIFIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kushang Patel, Research Associate Professor: School of Medicine: Anesthesiology and Pain Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007302; R01AG060992 (NIH)
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Osteo Arthritis Knee
Keywords: Osteoarthritis; chronic pain; behavioral health; exercise; physical activity; older adults
MeSH Terms: conditions — Osteoarthritis; Chronic Pain; Motor Activity | interventions — Behavioral Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral Health (Experimental): Ten behavioral health classes.
  Interventions: Behavioral: Behavioral Health
- Health Education (Active Comparator): Ten health education classes covering healthy aging.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Behavioral Health — Ten, group-based classes lasting one hour each that teaches symptom management and promotes physical activity.
  Arms: Behavioral Health
Behavioral: Health Education — Ten, group-based classes lasting one hour each that teaches topics related to aging and health (e.g., blood pressure control, maintaining healthy bones, cancer screening, immunizations).
  Arms: Health Education

SUMMARY:
This clinical trial will determine the added benefit of combining exercise and behavioral health education (versus exercise and aging and health education) to improve physical activity in community-dwelling older adults who have painful knee osteoarthritis (OA).

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a highly prevalent, leading cause of pain that limits physical functioning in older adults. Although clinical practice guidelines recommend physical exercise for managing symptoms of knee OA, several systematic reviews indicate that exercise intervention studies provide only short-term benefits (lasting 6 months) for knee OA. Many older adults with painful knee OA return to sedentary lifestyles when structured exercise programs end6. Efforts to increase and sustain physical activity in this population will require promoting self-regulatory skills to develop confidence to maintain an active lifestyle and manage symptoms that often limit activity. Therefore, we developed a group-based behavioral health (BH) program for older adults with painful knee OA that complements Enhance Fitness (EF) - a multicomponent, community-based exercise program for older adults, involving balance, strength, and endurance training. The Behavioral Health (BH) program will have 10, 1-hour weekly classes spread over 4 months, while the Health Education (HE) program will be equally matched for attention with classes on aging and health. In parallel with BH/HE programs, all study subjects will participate in Enhance Fitness (EF) exercise classes that will be held for 1-hour, 3 times a week for 4 months. EF+BH intervention (versus EF+HE) improves physical activity, pain, physical function, and other outcomes in older adults with knee OA. Due to the COVID-19 pandemic, all interventions transitioned to remote delivery in 2020.

ELIGIBILITY:
Inclusion criteria:

* Age 65 years or older
* Community-dwelling
* Physician diagnosis of knee OA
* Knee pain that occurs almost daily for at least the past 3 months
* Knee pain-related difficulty with walking or climbing stairs
* Stiffness in the knee for <30 min/day in the morning
* Crepitus in the knee

Exclusion criteria:

* Non-English speaking
* Cognitive impairment (Mini-Cog score ≤3)
* Unable or unwilling to give informed consent or accept randomization in either study group
* Unwilling to wear a thigh-mounted accelerometer for 1 week
* Significant, non-corrected visual or hearing impairment
* Plans to move out of the area in the next 12 months
* Plans to have knee, hip, or any other major surgery (including joint replacement) in the next 12 months
* Unable to walk a quarter of a mile independently (use of a straight cane is acceptable)
* Prior participation in cognitive-behavioral therapy or counseling for pain
* Exercises regularly (≥20 minutes/week of walking, hiking, dancing, or strength training, or participate in water exercise)
* Temporary exclusion: Any of the following in the past 6 months: cancer requiring treatment (except for non-melanoma skin cancer), heart attack or failure, stroke, hip fracture, hip/knee replacement, spinal surgery, heart surgery, deep vein thrombosis, or pulmonary embolus
* Temporary exclusion: Hospitalization in the past month
* Temporary exclusion: Currently undergoing physical therapy or rehabilitation treatment for knee OA or impairments in mobility function

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Average Number of Steps per day | 4 months,10 months
  Participant's average number of steps per day will be measured by a thigh mounted accelerometer (acitvPAL) worn for 1 week.

SECONDARY OUTCOMES:
Knee Pain and Function | 4 months, 10 months
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire will be used. This is a reliable, validated, and widely used patient-reported outcome measure for assessing knee pain and knee pain-related functional limitations in clinical trials of exercise in adults with knee OA. The knee pain and knee pain-related functional limitation subscales range 0-100 with higher scores indicating better outcome.
6 Minute Walk Test | 4 months, 10 months
  Mobility will be measured by the 6-Minute Walk Test. This is a recommended performance-based measures to assess interventions in adults with knee OA and in older adults in general, facilitating comparisons with previous exercise trials.
Timed Up and Go Test | 4 months, 10 months
  Mobility will be measured by the Timed up Go. This is a recommended performance-based measures to assess interventions in adults with knee OA and in older adults in general, facilitating comparisons with previous exercise trials.
Short Physical Performance Battery | 4 months, 10 months
  Mobility will be measured by the Short Physical Performance Battery. This is a recommended performance-based measures to assess interventions in adults with knee OA and in older adults in general, facilitating comparisons with previous exercise trials.
Fatigue | 4 months, 10 months
  The PROMIS-57 Profile v2.1 will be collected, which includes 8 question items on fatigue. The PROMIS fatigue score ranges 0-100 with higher scores indicating worse outcome.
Study Specific Treatment Satisfaction Questionnaire | 4 months, 10 months
  This multi-item measure assesses overall participant satisfaction with the study as well as individual treatment components. These questions were developed specifically for the PACIFIC Study. Overall and treatment-specific satisfaction scores range 20-100 with higher scores indicating better outcome.
Patient Global Impression of Change | 4 months, 10 months
  This is a widely used single item assessment of overall change in health status following treatment on a 7-point scale. Participants are asked, "Since the start of the study my overall status is: (1) Very much improved; (2) Much improved; (3) Minimally improved; (4) No change; (5) Minimally worse; (6) Much worse; and (7) Very much worse".

CONTACTS AND LOCATIONS:
Overall Officials: Kushang V Patel, PhD MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deshpande BR, Katz JN, Solomon DH, Yelin EH, Hunter DJ, Messier SP, Suter LG, Losina E. Number of Persons With Symptomatic Knee Osteoarthritis in the US: Impact of Race and Ethnicity, Age, Sex, and Obesity. Arthritis Care Res (Hoboken). 2016 Dec;68(12):1743-1750. doi: 10.1002/acr.22897. Epub 2016 Nov 3. PMID 27014966
- [Background] Leveille SG, Fried LP, McMullen W, Guralnik JM. Advancing the taxonomy of disability in older adults. J Gerontol A Biol Sci Med Sci. 2004 Jan;59(1):86-93. doi: 10.1093/gerona/59.1.m86. PMID 14718492
- [Background] Nelson AE, Allen KD, Golightly YM, Goode AP, Jordan JM. A systematic review of recommendations and guidelines for the management of osteoarthritis: The chronic osteoarthritis management initiative of the U.S. bone and joint initiative. Semin Arthritis Rheum. 2014 Jun;43(6):701-12. doi: 10.1016/j.semarthrit.2013.11.012. Epub 2013 Dec 4. PMID 24387819
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee. Cochrane Database Syst Rev. 2015 Jan 9;1(1):CD004376. doi: 10.1002/14651858.CD004376.pub3. PMID 25569281
- [Background] Newberry SJ, FitzGerald J, SooHoo NF, Booth M, Marks J, Motala A, Apaydin E, Chen C, Raaen L, Shanman R, Shekelle PG. Treatment of Osteoarthritis of the Knee: An Update Review [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2017 May. Report No.: 17-EHC011-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK447543/ PMID 28825779
- [Background] Focht BC. Effectiveness of exercise interventions in reducing pain symptoms among older adults with knee osteoarthritis: a review. J Aging Phys Act. 2006 Apr;14(2):212-35. doi: 10.1123/japa.14.2.212. PMID 19462551
- [Background] Newman AB, Bayles CM, Milas CN, McTigue K, Williams K, Robare JF, Taylor CA, Albert SM, Kuller LH. The 10 keys to healthy aging: findings from an innovative prevention program in the community. J Aging Health. 2010 Aug;22(5):547-66. doi: 10.1177/0898264310363772. Epub 2010 May 21. PMID 20495156